CLINICAL TRIAL: NCT06823063
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of a Single Dose of Human Umbilical Cord Mesenchymal Stem Cell Injection (IxCell hUC-MSC-P) in Patients With Connective Tissue Disease-associated Interstitial Lung Disease
Brief Title: Clinical Trial of Human Umbilical Cord Mesenchymal Stem Cells (IxCell hUC-MSC-P) in the Treatment of CTD-ILD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai IxCell Biotechnology Co., LTD (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC-MSC-ILD21003
Record Dates: First submitted 2025-01-14; First posted 2025-02-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: CTD-ILD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hMSCs 5.0×10^7 (Experimental): Human umbilical cord mesenchymal stem cells（hMSCs）5.0×10^7 cells
  Interventions: Biological: MSC
- hMSCs 10.0×10^7 (Experimental): Human umbilical cord mesenchymal stem cells（hMSCs）10.0×10^7 cells
  Interventions: Biological: MSC
- hMSCs 20.0×10^7 (Experimental): Human umbilical cord mesenchymal stem cells（hMSCs）20.0×10^7 cells
  Interventions: Biological: MSC

INTERVENTIONS:
Biological: MSC — a single injection dose i.v.

SUMMARY:
To evaluate the safety and tolerability of IxCell hUC-MSC-P in the treatment of patients with connective tissue disease-related interstitial lung disease.

To evaluate the efficacy, pharmacokinetics and immunogenicity of IxCell hUC-MSC-P in the treatment of connective tissue disease-associated interstitial lung disease (CTD-ILD).

DETAILED DESCRIPTION:
Mesenchymal stem cells (MSCs) are a kind of adult stem cells, which express CD73, CD40 and CD105 on the cell surface, but not CD34, CD45 and HLA-DR. They can self-renew in vitro culture environment and have the ability to differentiate into bone, adipose and chondrocytes.

Because of its anti-inflammatory, immunomodulatory and natural regenerative functions, it has become a potential therapeutic drug to control lung immune dysfunction and inflammatory response. MSCs can regulate the microenvironment of injured tissues by secreting anti-inflammatory factors and exert immunomodulatory ability through cell interaction. Firstly, MSCs can directly inhibit the proliferation of T cells, thereby reducing the number of T cells in the inflammatory site. Secondly, MSCs can also suppress T cell responses through paracrine effects. MSCs can secrete soluble immunosuppressive factors such as prostaglandin E2 (PEG2), transforming growth factor β (TGF-β), indole2, 3-dioxygenase (IDO) and nitric oxide (NO) to inhibit the ongoing T cell inflammatory response and promote T cell apoptosis. Thirdly, MSCs can attenuate the antigen-presenting ability of dendritic cells (DCs) by inhibiting DCS; Fourth, MSC-induced DCs showed a tolerogenic phenotype, which promoted the transformation of inflammatory M1 macrophages into immunosuppressive M2 macrophages. Fifth, in the manner described above, MSCs reduce the production of inflammatory factors (TNF-α, IL-1β, and IL-12) in DC cells and M1 macrophages, promote the production of anti-inflammatory factors IL-10 and TGF-β, and promote tissue repair and regeneration capacity. At the same time, immunotolerant DCs and M2 macrophages induce MSCs to produce human leukocyte antigen (HLA) G5, which promotes MSCS-induced Treg cells to form an anti-immune environment around the injured lung tissue.

The development of CTD-ILD is accompanied by chronic inflammation, and the use of MSCs can alleviate this inflammatory response. Some animal experiments and in vitro culture studies have also shown that MSCs can differentiate into alveolar epithelial cells and have potential regenerative treatment ability for lung diseases. By routine intravenous infusion, MSCs can be captured by the pulmonary vasculature and facilitate the treatment of lung injury. According to the above immunomodulatory and anti-inflammatory functions of MSCs, MSCs therapy can theoretically inhibit the inflammatory response of CTD-ILD and block or even reverse the process of pulmonary fibrosis in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes, aged 18-80 years;
2. SSc diagnosed according to the 2013 American College of Rheumatology and European League Against Rheumatism (ACR/EULA) criteria:
3. Pulmonary fibrosis ≥10% was confirmed by high-resolution chest computed tomography (HRCT);
4. The diffusion capacity for carbon monoxide (DLco) was 30%-89% of the expected value, and progression of interstitial lung disease was found. Progression was confirmed if one of the following criteria was met:

   1. A decline of 10% or more in the percentage of predicted forced vital capacity (FVC%p) within 24 months (significant decline in ventilatory function) despite treatment;
   2. A decline of ≥5% in FVC%p + a decline of ≥15% in DLco (a decline in ventilation function + a decline in diffusion capacity) within 24 months despite treatment;
   3. Within 24 months, high resolution CT (HRCT) showed worsening of pulmonary fibrosis + ≥5% decline in FVC%p (deterioration of lung imaging + decline in ventilatory function), despite treatment.
   4. Despite the treatment, 24 months reduced FVC % p + 5% or higher clinical symptoms (reduced ventilation function + symptoms);
   5. Worsening of pulmonary fibrosis on HRCT + worsening of clinical symptoms (worsening of lung imaging + worsening of symptoms) within 24 months despite treatment;
5. Forced Vital Capacity (FVC) was greater than 40% of expected vital capacity;
6. The patient was able to complete the 6-Minute Walk Test (6MWT);
7. Be able to understand and complete pulmonary function test procedures.
8. Fully informed experiment purposes, methods, and possible uncomfortable, willing to medicine and follow-up inspection on time, according to the requirements of plan agreed to participate in trials, and sign the informed consent.

Exclusion Criteria:

1. The patients were diagnosed with other lung diseases other than SSc-ILD, such as COPD, lung abscess, lung cancer and other types of connective tissue disease-related interstitial lung disease.
2. Have obvious acute lung infection requiring anti-infection treatment (treatment of 4 weeks prior to the start of the respiratory tract infection and systemic infection);
3. History of severe pulmonary hypertension, including right heart failure, cardiac intubation, and parenteral administration of prostaglandin analogues;
4. History of myocardial infarction or angina pectoris within 6 months before enrollment;
5. Patients with 3 or more fingertip ulcers when signing the informed consent form or unable to accurately observe fingertip ulcers due to other reasons of the hand;
6. Allergic to any component of the medication;
7. Life expectancy of less than 1 year due to diseases other than SSc;
8. Planned surgical procedures during the trial;
9. Has a history of scleroderma kidney crisis;
10. Patients who had used glucocorticoids within 2 weeks before enrollment but could not maintain the dosage ≤10mg/ d equivalent prednisone;
11. Patients who had used methotrexate within 2 months before enrollment, or failed to maintain a stable dosage while using other immunosuppressants;
12. Into groups of 2 months before used anti fibrosis drug (such as pyrazole ketone, dani, cloth, etc.);
13. Patients treated with rituximab, tocilizumab and mesenchymal stem cells within 2 months before enrollment;
14. Patients with other systemic diseases and organ dysfunction (ALT>1.5 times upper limit of normal; Cr>1.5 times upper limit of normal; LVEF≤40%; Other progressive or uncontrolled diseases);
15. Active hepatitis, tuberculosis, HIV infection;
16. Patients with malignant tumors or a history of cancer;
17. Pregnant or lactating women or those who have recently planned to have children and cannot take effective contraceptive measures;
18. People with a history of alcohol or drug abuse;
19. Enrolled in another drug trial within 3 months before enrollment;
20. Unable to complete all assessors;
21. And anyone who was deemed by the investigator to be ineligible for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AE | 1 week, 2 weeks, 4 weeks, 12 weeks, 24 weeks
  Adverse events and serious adverse events.
Forced Vital Capacity（FVC） | 24 weeks
  Absolute change in FVC

SECONDARY OUTCOMES:
Forced Expiratory Volume in One Second (FEV1) | 12 weeks, 24 weeks
  Forced expiratory volume in 1 second (FEV1)
Diffusing Capacity of the Lung for Carbon Monoxide (DLco) | 12 weeks, 24 weeks
  Absolute change in carbon monoxide diffusing capacity (DLco)
St. George's Respiratory Questionnaire (SGRQ） | 12 weeks, 24 weeks
  Score range: 0-100； Higher scores indicate worse health status, while lower scores indicate better health； Changes in the St George's Respiratory questionnaire (SGRQ)
Short Form Health Survey (SF-36) | 12 weeks, 24 weeks
  Score range: 0-100； Higher scores indicate better health status, while lower scores indicate worse health； Changes in the Short Form Health Survey (SF-36)；
Modified Rodnan Skin Score(MRSS) | 12 weeks, 24 weeks
  Score range: 0-51； Higher scores indicate worse health status, while lower scores indicate better health； Changes in the modified Rodnan Skin Score (MRSS)
High-resolution computed tomography (HRCT) | 12 weeks, 24 weeks
  Pulmonary interstitial fibrosis on high-resolution computed tomography (HRCT)
6-MWT | 12 weeks, 24 weeks
  Changes of oxygen saturation and walking distance in six-minute walk test (6MWT)
Health assessment questionnaire (HAQ) | 12 weeks, 24 weeks
  Score range: 0-3； Higher scores indicate worse health status, while lower scores indicate better health； Changes in health assessment questionnaire (HAQ)
Survival | 12 weeks, 24 weeks
  Disease progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: tao Ren, Doctor, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China